CLINICAL TRIAL: NCT07123597
Title: Effect of Thickness Variation in Coronal Plug on Root Maturation and Periapical Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rania ElSayed Soliman (Other)
Collaborators: Benha National University (Other)
Responsible Party: Sponsor-Investigator, Rania ElSayed Soliman, assistant lecturer, Benha National University
Organization: Benha National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Regenerative Endodontics
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Immature Permanent Teeth With Open Apex
Keywords: regenerative endodontics; root maturation; periapical healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: Teeth will be treated by regenerative endodontic procedures with placing of 5mm coronal plug.
  Interventions: Other: 5mm bioceramic putty coronal plug
- Group B (Experimental): Group B: Teeth will be treated by regenerative endodontic procedures with placing of 3mm coronal plug.
  Interventions: Other: 3mm bioceramic putty coronal plug

INTERVENTIONS:
Other: 5mm bioceramic putty coronal plug — Teeth will be treated by regenerative endodontic procedures with placing of 5mm bioceramic putty coronal plug.
  Arms: Group A
Other: 3mm bioceramic putty coronal plug — Teeth will be treated by regenerative endodontic procedures with placing of 3mm bioceramic putty coronal plug.
  Arms: Group B

SUMMARY:
d. Second visit:

After 3 weeks the patients will be randomly divided into 2 groups:

Group A:

Patients will be anesthetized 1 carpule of mepivacaine without vasoconstrictor (Mepivacaine HCl 3%), the access will be reopened under rubber dam isolation and the canal will be irrigated with a total of 20 ml of 1.5-2.5% sodium hypochlorite solution. The canal will then be dried with sterile paper points; a sterile sharp needle will be used to irritate the apical tissue until bleeding occurred apically in the root canal space so as to create a biological scaffold for the regenerative process.

Over a 15-minute time period, the blood will be allowed to clot to a level of 3 mm below the cemento-enamel junction. A resorbable matrix such as CollaPlug™, Collacote™, CollaTape™ will be placed over the blood clot if necessary. Then 3 mm of MTA will be placed using a suitable size amalgam carrier. A damped cotton pellet on a tweezer placed above the unset MTA and large condenser will be used to seal the canal orifice completely. The access cavity will be sealed with Fuji IX glass ionomer filling material and acid etched composite resin bonded filling material.

Group B:

The same procedures that will be followed in group A will be also done in group B, except for the thickness of MTA coronal plug which will be 5mm in its thickness

e. Follow-up:

The patients will be recalled after 1, 6 and 12 months for follow up. The post-treatment follow-up examination will be accomplished as follows:

* CBCT scan will be done at 6 and 12 months follow up appointments.
* An evaluation was performed on each patient to assess presence of any signs and symptoms clinically by inspection, percussion, palpation, or biting on the treated tooth.

DETAILED DESCRIPTION:
4.1. Trial Design: The trial design of this study is a prospective, 2-arm, 1:1, parallel, randomized, clinical trial (RCT). In RCT, participants are allocated at random to receive one of several interventions according to the research plan created by the investigators. These interventions may be drug, placebo or certain procedure which is not usually known whether it will be helpful, harmful or with no difference than the available alternatives. In RCT the outcomes are measured, so it is considered a quantitative study. This trial design methodology conforms to the Consolidated Standard of Reporting Trials (CONSORT).

4.2. Participants:

a. Sample size: Teen participants will be selected from the out patients of the endodontic clinic Faculty of dentistry, Ain Shams University), 9 cases in each group .

4.3. Randomization: Randomization is a process that assigns research participants by chance, rather than by choice, to either the experimental group or the control group. The goal of randomization is to produce comparable groups in terms of general participant characteristics, such as age, gender, chief complain, time pass after trauma, and the other key factors that affect the probable course the disease would take. In this way, the 2 groups are as similar as possible at the start of the study. At the end of the study, if one group has better outcome than the other, the investigators would be able to conclude with some confidence that one intervention is better than the other.

Randomization process was achieved in three steps:

1. Sequence generation:

   Sequence generation will be done for the patient's number (from 1 to 10) using computer sequence generation (www.random.org) which will give a table for group A and group B with randomized patient's numbers (5 number in each group).
2. Allocation concealment mechanism:

   It is a procedure for protecting the randomization process so that the treatment to be allocated is not known before the patient participated in the study. For the allocation concealment mechanism, each of 10 papers (each paper was eight folded) numbered from 1 to 10 were, individually packed, in opaque envelopes. Each participant picked an envelope at the beginning of the second visit. The number in the envelope determined which procedure will be performed to the patient. The partner will decide the procedure for the operator according to that number.
3. Implementation:

The random allocation sequence will be done in the Center of The Evidence Based Dentistry, Faculty of Oral and Dental Medicine, Ain Shams University. However, allocation concealment and participant assignment to the intervention will be done by the other investigator.

4.4. Blinding (Masking): Double blinded (Patient and Assessor). Patient will not informed what procedure he/she was subjected to. Assessor will be blinded to the intervention applied on the patient (during pain and swelling assessment).

4.5. Intervention:

Preoperative CBCT scan:

A preoperative CBCT scan will be done to all cases with a high resolution Cone Beam Computed Tomography machine (Planmeca ProMax 3d MID; Planmeca, Helsinki, Finland), with endodontic mode, operating at 90 KV, 12mA with a voxel dimension of 75μm.

In this study 18 patients will be randomly divided into 2 groups (9 patients per each group), where treatment will be completed in 2 visits.

First visit:

A calcium hydroxide intracanal medicament will be utilized in all teeth of both groups.

Second visit:

Group A: Teeth will be treated by regenerative endodontic procedures with placing of 3mm MTA coronal plug .

Group B: Teeth will be treated by regenerative endodontic procedures with placing of 5mm MTA coronal plug.

ELIGIBILITY:
Inclusion Criteria:

* All patients were medically free [American Society of Anesthesiologists (ASA) Class I or II].
* Age ranging between 10-18 years old.
* No sex predilection.
* Patients having asymptomatic and/or symptomatic immature necrotic anterior teeth.

Exclusion Criteria:

* Patients with a history of allergy to any of the material used in the study.
* Patients with systemic diseases (e.g. diabetes mellitus, bleeding disorders, heart diseases, liver diseases, kidney diseases, genetic disorders and syndromes).
* Psychologically disturbed patients.
* Teeth that needed a post and core as the final restoration.
* Patients who had teeth with periodontal pockets more than 3 mm or generalized chronic periodontitis
* Teeth with developmental anomalies (i.e., dens invaginatus or a palatogingival groove)
* Patients who had radiographic evidence of external / internal root resorption or cystic lesion.
* Patients refused participating in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Root maturation | after 12 month
  after superimposition of the pre and post operative CBCT percentage growth of the root was calculated after
  1. measuring the root length in millimeter in the pre and post operative CBCT increase in length = (follow up length - base line length).
  2. Amount of radiographic increase in the root dentinal wall thickness Dentin thickness in the post operative CBCT = (root thickness-pulp space) and was compared to the baseline CBCT radiograph.
     The increase in thickness was calculated as follows: increase in thickness = (follow-up thickness -base line thickness).
  3. measuring the decrease of apical diameter: Using the preset measurement scale, the diameter of the apical foramen was measured in millimeters on the 12 months follow up CBCT radiograph and was compared to the baseline CBCT radiograph (decrease of apical diameter = follow-up apical diameter-base line apical diameter).

SECONDARY OUTCOMES:
periapical healing | 12 month
  1. Clinically: By visual inspection of the patient's soft tissue at 1, 3, 6 and 12 months (Swelling). When the case is symptoms-free, i.e., without sinus tract swelling, pain on palpation, or percussions, the case is considered a success.
  2. Radiographically:
  Measuring of the total lesion volume on the 12 months follow up CBCT radiograph and compared to the baseline CBCT radiograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha National University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
photographs, radiographs, age, sex, general health condition
Supporting Information: Study Protocol